CLINICAL TRIAL: NCT03119558
Title: 18F-Florbetaben (Neuraceq®) PET/MRI Evaluation of Cardiac Amyloid
Brief Title: PET/MRI Evaluation of Cardiac Amyloid
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology - Nuclear Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35049
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Florbetaben (Neuraceq®) PET/MRI (Experimental): Participants with known or suspected cardiac amyloidosis will be injected with 8 mCi of 18F-Florbetaben (Neuraceq®) and undergo the PET/MRI image acquisition 45-60 minute post-injection. PET and MRI data will be acquired simultaneously to ensure optimal timing and spatial correspondence between MRI and PET data. Total scan time will take approximately 60 minutes.
  Interventions: Drug: 18F-Florbetaben (Neuraceq®) PET/MRI

INTERVENTIONS:
Drug: 18F-Florbetaben (Neuraceq®) PET/MRI — Administration of 8.0 mCi 18F-Florbetaben (Neuraceq®) IV followed by simultaneous acquisition PET emission and cardiac MRI sequence scan 45-60 minutes post-injection.

SUMMARY:
Cardiac amyloidosis is a disorder characterized by the deposition of abnormal proteins called amyloid in the heart tissue. This makes it difficult for the heart to function properly. The investigators wish to evaluate if the radiopharmaceutical 18F-Florbetaben (Neuraceq®) that targets beta amyloid can also identify cardiac amyloid deposition.

DETAILED DESCRIPTION:
The use of hybrid positron emission tomography/ magnetic resonance imaging (PET/MRI) scanners in clinical practice enhance the ability to evaluate the heart from both an anatomical and functional perspective. It is hypothesized that an increased PET signal of 18F-Florbetaben (Neuraceq®) will be detected in cardiac amyloid deposits within the heart tissue, while the MRI provides the anatomical information. The ability to reliably and non-invasively image amyloid deposition in the heart would be potentially advantageous in the following scenarios:

1. Diagnosis of cardiac amyloidosis
2. Decreasing unnecessary invasive myocardial procedures.

The investigators believe this trial will help expand the use of current PET amyloid tracers and help many patients who currently undergo myocardial biopsy for the diagnosis of cardiac amyloid.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the scan
* Patient with known or suspected cardiac amyloidosis.
* Patient is capable of complying with study procedures

Exclusion Criteria:

* Patient is pregnant or nursing
* Metallic implants (contraindicated for MRI)
* History of renal insufficiency (only for MRI contrast administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with 18F-Florbetaben (Neuraceq®) uptake on Fused PET/MRI Images | an estimated average of 2 hours
  Diffuse (widespread), focal (point) and focal-on-diffuse (combination of the two) patterns of 18F-Florbetaben uptake will be considered positive findings indicating cardiac amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baratto L, Park SY, Hatami N, Gulaka P, Vasanawala S, Yohannan TK, Herfkens R, Witteles R, Iagaru A. 18F-florbetaben whole-body PET/MRI for evaluation of systemic amyloid deposition. EJNMMI Res. 2018 Jul 24;8(1):66. doi: 10.1186/s13550-018-0425-1. PMID 30043115